CLINICAL TRIAL: NCT01247662
Title: Psychometric Studies of the Chinese Versions of the Social Responsiveness Scale, the Childhood Asperger's Syndrome Test, and the Autism Spectrum Quotient
Brief Title: Psychometric Studies of the Chinese Versions of the SRS, CAST, and AQ
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201005041R
Record Dates: First submitted 2010-11-22; First posted 2010-11-24 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2012-04

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism spectrum disorder; Social Responsiveness Scale; Childhood Asperger's Syndrome Test; Adult Autism Spectrum Quotient; psychometric
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- ASD group
- ADHD group
- Normally developing control group

SUMMARY:
Autism spectrum disorder (ASD) is a pervasive neurodevelopmental disorder with prominent reciprocal social and communication impairment and restricted repetitive behavior or interest. ASD is a highly heritable disease with tremendous impact on individuals, families, and society. In addition to the interview instruments, self-administered rating scales are commonly used in screening, assessment of symptoms' change, and evaluation of intervention effects. The Social Responsiveness Scale, the Childhood Asperger's Syndrome Test, and the Autism Spectrum Quotient are internationally widely used rating scales measuring autistic traits in both clinical and community samples in western counties. Establishment of internationally-recognized reliable and valid instruments is not only useful for clinical screening, but also helpful in future functional outcomes, neurocognitive, genetic and brain imaging studies.

DETAILED DESCRIPTION:
Specific Aims:

1. To identify the factor structures and norms of the SRS, CAST, and AQ;
2. To assess the concurrent validity of the SRS, CAST, and AQ;
3. To assess the discriminative validity of the three scales by testing the difference of total scores and subscales scores of the SRS, CAST, and AQ between the ASD, attention-deficit hyperactivity disorder (ADHD), and control groups;
4. To correlate the autistic characteristics between parents and children and compare the magnitude of correlations of autistic traits across the 3 groups.

This is a cross-sectional questionnaire survey in school-based and clinic-based samples. The participants include (1) ASD group: 200 cases with DSM-IV ASD; (2) ADHD group: 200 cases with DSM-IV ADHD; (3) Normally developing control group: a school-based sample of around 1200 grade 1 to grade 8 students. 100 students randomly selected from school-based sample will be reassessed at a 2-week interval for the test-retest reliability study. The teachers will complete the SRS and SNAP-IV (for ADHD symptoms); parents will report on their children on the SCQ, SRS, CAST, SNAP-IV, and CBCL, and report themselves on the SRS, AQ, and ASRI; children will report on themselves using the SRS, AQ, SNAP-IV, and YSR. Parents of clinical participants will be interviewed by the ADI-R or K-SADS-E to confirm their diagnosis of ASD and ADHD, respectively.

We expect that this study will reach the following objectives:

1. To establish psychometric properties of the Chinese versions of SRS, CAST, and AQ for future use in clinical, school, and research settings;
2. To obtain the preliminary information about the prevalence of ASD, and understand the correlation of autistic traits in family;
3. To enhance the awareness of school teachers and counselors about ASD among students.

ELIGIBILITY:
Inclusion Criteria:

* Control group: Subjects without ADHD or ASD;
* ADHD group & ASD group: subjects have a clinical diagnosis of ADHD, or ASD defined by the Diagnostic and Statistical Manual, Fourth Edition (DSM-IV), which was made by a full-time board-certificated child psychiatrist at the first visit and following visits.

Exclusion Criteria:

* The subjects will be excluded from the study if they currently meet criteria or have a history of the following condition as defined by DSM-IV: Schizophrenia, Schizoaffective Disorder, Organic Psychosis, Mental Retardation, or Pervasive Developmental Disorder. Moreover, the subjects will be excluded from the control group if have a history of the following condition as defined by DSM-IV: ADHD or ASD in addition to the above exclusion criteria.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The participants include (1) ASD group: 200 cases with DSM-IV ASD; (2) ADHD group: 200 cases with DSM-IV ADHD; (3) Normally developing control group: a school-based sample of around 1200 grade 1 to grade 8 students.
Sampling Method: Non-Probability Sample
Enrollment: 2460 (Actual)
Dates: Start 2011-01; Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shur-Fen Gau, MD, PhD, Principal Investigator — National Taiwan University Hospital & College of Medicine
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan